CLINICAL TRIAL: NCT03159845
Title: A Mono-centric, No-profit, Case-control Study With Daily Oral Supplementation of Zinc Sulphate After Autologous Stem Cell Transplantation in Patients Affected by Multiple Myeloma
Brief Title: Zinc as Enhancer in Immune Recovery After Stem Cell Transplantation for Hematological Malignancies
Acronym: ZENITH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Lorenzo Iovino, MD, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hematology AOUPisa
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stem Cell Transplant Complications
Keywords: zinc
MeSH Terms: interventions — Levofloxacin; Tablets; Fluconazole; Acyclovir

STUDY DESIGN:
Intervention Model Description: Case-control study, open, without placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): patients undergone autologous stem cell transplantation. They take levofloxacin 500 mg/d, aciclovir 400 mg bid, fluconazole 200 mg bid from day +10 until day +30 after stem cell transplantation
  Interventions: Drug: Levofloxacin 500Mg Oral Tablet; Drug: Fluconazole 200mg tab; Drug: Acyclovir 400 MG
- Zinc (Experimental): patients undergone autologous stem cell transplantation. They take the same antimicrobial prophylaxis of patients of the Control group, and, in addition, a daily oral supplementation of Zinc Sulfate, 600 mg/die, uncoated tabs, from day +5 until day +100 after transplant
  Interventions: Drug: Zinc Sulfate Oral Product; Drug: Levofloxacin 500Mg Oral Tablet; Drug: Fluconazole 200mg tab; Drug: Acyclovir 400 MG

INTERVENTIONS:
Drug: Zinc Sulfate Oral Product
  Arms: Zinc
Drug: Levofloxacin 500Mg Oral Tablet — once daily from day +10 until day +30 after stem cell transplantation
Drug: Fluconazole 200mg tab — twice daily from day +10 until day +30 after stem cell transplantation
Drug: Acyclovir 400 MG — twice daily from day +10 until day +30 after stem cell transplantation

SUMMARY:
Patients affected by multiple myeloma undergone autologous stem cell transplantation (SCT) are enrolled at the moment of stem cell collection. They are randomized 1:1 in two groups at the moment of the graft. Patients of the Control group take only standard antimicrobial prophylaxis after SCT; the Sample group takes in addition a daily oral supplementation of Zinc Sulfate (600 mg/die) from day +5 until day +100 after SCT. Laboratory tests are performed on peripheral blood samples.

DETAILED DESCRIPTION:
Patients affected by multiple myeloma undergone autologous stem cell transplantation (SCT) are enrolled at the moment of stem cell collection. They are randomized 1:1 in two groups at the moment of the graft. Patients of the Control group take only standard antimicrobial prophylaxis after SCT; the Sample group takes in addition a daily oral supplementation of Zinc Sulfate (600 mg/die) from day +5 until day +100 after SCT. The aim of the study is to investigate the immune reconstitution in presence of Zinc, focused on thymic reconstitution. Laboratory tests are performed on peripheral blood samples, collected at 4 time-points: two before transplant (at the moment of the enrollment and the day before conditioning) and two after transplant (day +30 and +100).

ELIGIBILITY:
Inclusion Criteria:

* eligibility to stem cell transplantation

Exclusion Criteria:

* allergy to Zinc
* copper deficiency or Wilson's syndrome
* patients who admit zinc assumption in other drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Thymic output improvement by TRECs | increase of TRECs levels from day +30 until day +100 after transplant
  Measure of T cell receptor excision circles levels on peripheral lymphocytes (TRECs), calculated as number of copies of TRECs/mcLin droplet digital PCR
Thymic output improvement by flow cytometry | days +30, +100 after transplant
  Measure of circulating T naive lymphocytes by 8-colour flow-cytometry. T naive are identified as CD4+/CD8+ lymphocytes with the coexpression of CD45RA, CD27, CD28. The value is estimated as number of T naive/mcL

SECONDARY OUTCOMES:
Variations in circulating lymphocyte populations | days +30, +100 after transplant
  Flow cytometry to determine the variations of t cell subpopulations after graft
Immune competence | days +30, +100 after transplant
  quantitative polymerase chain reaction on peripheral blood aiming to quantify Torquetenovirus viral load
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | days +30, +100 after transplant
  case report form to report side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology UO, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iovino L, Mazziotta F, Carulli G, Guerrini F, Morganti R, Mazzotti V, Maggi F, Macera L, Orciuolo E, Buda G, Benedetti E, Caracciolo F, Galimberti S, Pistello M, Petrini M. High-dose zinc oral supplementation after stem cell transplantation causes an increase of TRECs and CD4+ naive lymphocytes and prevents TTV reactivation. Leuk Res. 2018 Jul;70:20-24. doi: 10.1016/j.leukres.2018.04.016. Epub 2018 May 2. PMID 29747074